CLINICAL TRIAL: NCT06823986
Title: The Relation Between Extraction Space Consumption and Overjet Reduction During Maxillary Anterior En-Masse Retraction by Two Levels of Force Application
Brief Title: Extraction Space Consumption and Overjet Reduction After Maxillary Anterior Enmasse Retraction in Orthodontics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Omnia Megahed, Principal investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Extraction and retraction
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Extraction Space Consumption and Overjet Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retraction with mini screw and power arm (Experimental): Ten patients will be treated with mini screw and power arm
  Interventions: Device: Retraction of anterior teeth by putting miniscrews and power arm
- Retraction with mini screw and welded hook in main wire arch (Experimental): Ten patients will be treated with mini screw and welded hook in main wire arch
  Interventions: Device: Retraction of upper anterior teeth by putting miniscrews and welded hooks in main wire arch

INTERVENTIONS:
Device: Retraction of anterior teeth by putting miniscrews and power arm — Enmasse retraction of upper anterior teeth after extraction of upper first permanent premolar on miniscrews and power arm
  Arms: Retraction with mini screw and power arm
Device: Retraction of upper anterior teeth by putting miniscrews and welded hooks in main wire arch — Enmasse retraction of upper anterior teeth after extraction of upper first permanent premolars on miniscrews and welded hooks in main wire arch
  Arms: Retraction with mini screw and welded hook in main wire arch

SUMMARY:
Extraction space consumption and overjet reduction after maxillary anterior enmasse retraction in orthodontics

DETAILED DESCRIPTION:
The Relation between Extraction Space Consumption and Overjet Reduction during Maxillary Anterior En-Masse Retraction by Two Levels of Force Application

ELIGIBILITY:
Inclusion Criteria:

* 1. Young adult male and female patients (Age range from 18 to 25 years) with maxillary dental protrusion.

  2. Patients with Angle class I or class II division I malocclusion with maxillary anterior teeth protrusion and proclination. 3. Skeletal class I. 4. Healthy compliant and motivated patient. 5. No missing of any tooth except wisdom teeth. 6. Good oral hygiene.

Exclusion Criteria:

* 1. Previous orthodontic treatments. 2. Any systemic or bone diseases. 3. Pregnant and lactating patient. 4. Smoking history. 5. Presence of periodontal diseases. 6. Previous maxillary anterior surgery. 7. Gingival overgrowth.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
extraction space consumption and amount of overjet reduction in millimeters. | 2 years
  Cone beam computed tomography and cast scanning

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abdo Ibrahem, Professor, Principal Investigator — Professor of orthodontics
Locations (1):
- Omnia Megahed Hussein Hemeid, Cairo, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: No